CLINICAL TRIAL: NCT03120650
Title: Scalp Acupuncture for Dyskinesia After Ischemic Stroke
Acronym: LUSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LUS64385700
Record Dates: First submitted 2017-04-11; First posted 2017-04-19 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scalp acupuncture (Experimental): number:58 The needle will be maintained in place for 30 minutes. Patients in both groups will receive rehabilitation five times per week (Monday through Friday) for 8 consecutive weeks.
  Interventions: Other: Scalp acupuncture
- Conventional rehabilitation (Active Comparator): number:58 Rehabilitation will be conducted for 1 hour five times per week (Monday through Friday) for 8 weeks.
  Interventions: Other: Conventional rehabilitation

INTERVENTIONS:
Other: Scalp acupuncture — Acupoint selection: Shenting (DU24; Baihui (DU20; and upper 1/5 and middle 2/5 in the contralateral motor area (upper: 0.5 cm posterior to the midpoint of the front and rear midline; middle 2/5: intersection between the eyebrow line and the leading edge of the temple hairline.
  Arms: Scalp acupuncture
Other: Conventional rehabilitation — Rehabilitation plans will be made according to the Guidelines for Stroke Rehabilitation in China (Cerebrovascular Disease Association and the Neurological Rehabilitation Association of Neurology Branch of the Chinese Medical Association, 2012), including physical therapy and occupational therapy.
  Arms: Conventional rehabilitation

SUMMARY:
Scalp acupuncture formed by combining traditional Chinese acupuncture techniques and modern theories in medical anatomy has been widely used to treat ischemic stroke in China, but effective clinical trials that verify its efficacy are lacking. This study proposes to verify the effects of Lu's scalp acupuncture on ischemic stroke by comparing differential improvement of motor function between conventional rehabilitation alone and conventional rehabilitation with Lu's scalp acupuncture.

DETAILED DESCRIPTION:
A randomized, controlled, parallel, clinical trial. 116 ischemic stroke patients will be collected with dyskinesia from Longhua Hospital, Shanghai University of Traditional Chinese Medicine and Huashan Hospital, Fudan University in China. All patients will be equally randomized into either a control group (conventional rehabilitation) or an experimental group (scalp acupuncture + conventional rehabilitation). In the control group, patients will receive conventional rehabilitation according to the Guidelines for Stroke Rehabilitation in China. In the experimental group, conventional rehabilitation will be supplemented with oblique acupuncture at approximately 15° and an insertion depth of 25-35 mm in the motor areas of the scalp. Twisting speed will be 200 times per minute. Acupuncture will be performed six times per day in 1-minute bouts, with a 4-minute rest following each bout. Patients in both groups will receive rehabilitation five times per week for 8 consecutive weeks. The primary outcome will be the difference in Fugl-Meyer motor function score between posttreatment (4 weeks, 8 weeks, and 6 months of follow-up) and baseline.

The secondary outcomes will be differences in the Modified Barthel Index, stroke-specific quality of life, and stroke syndrome of traditional Chinese medicine.

ELIGIBILITY:
Inclusion Criteria:

* Meet to criteria for diagnosis and efficacy evaluation of stroke, formulated by The State Administration of Traditional Chinese Medicine Encephalopathy Emergency Cooperative Group in 1996 (trial implementation)

  * Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke in China in 2014 (Neurology Branch of Chinese Medical Association and Cerebrovascular Disease Association of Neurology Branch of Chinese Medical Association, 2015)
  * Ischemic stroke diagnosed by CT or magnetic resonance imaging (MRI), with the presence of stable vital signs and awareness
  * An age of 40-70 years Onset within 1-6 months
  * Motor dysfunction in the extremities
  * A Mini-Mental State Examination (Pangman et al., 2000) score > 24 points

Exclusion Criteria:

* Consciousness disorder or severe cognitive impairment

  * Severe Parkinson's disease, heart disease, cancer, epilepsy, or chronic alcoholism
  * Hepatic or renal impairment
  * Hemorrhagic tendency
  * Sensitivity to acupuncture
  * Congenital disability
  * Pregnancy
  * Currently participating in other clinical trials

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2023-03-20 (Estimated)

PRIMARY OUTCOMES:
The Fugl-Meyer Assessment (FMA) | 8 week
  Fugl-Meyer motor function score can effectively assess the degree of dyskinesia at different times during recovery after stroke.

SECONDARY OUTCOMES:
The Fugl-Meyer Assessment (FMA) | 16 week
  Fugl-Meyer motor function score can effectively assess the degree of dyskinesia at different times during recovery after stroke.
modified Barthel Index (mBI) | 8 week, 16 week
  to evaluate the daily life function, including stool, urine, dressing, using the toilet, eating, transfer, walking for 45 meters, wearing clothes, going up and down stairs, and bathing.
Stroke syndrome of traditional Chinese medicine (SSTCM) | 8 week, 16 week
  self-rating scale that reflects the quality of life of stroke patients
fractional amplitude of low frequency fluctuation (fALFF) | 8 week
  fALFF aquired by fMRI technique measures the relative contribution of low frequency ﬂuctuations within a speciﬁc frequency band to the whole detectable frequencyrange

CONTACTS AND LOCATIONS:
Overall Officials: jian, Study Director — Shanghai University of Traditional Chinese Medicine
Locations (2):
- China (2):
  - Longhua Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Longhua hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhan Y, Pei J, Wang J, Fu Q, Xu J, Yan M, Cai Y, Cui X, Ye W, Fan M, Yu Q, Jia J. Motor function and fALFF modulation in convalescent-period ischemic stroke patients after scalp acupuncture therapy: a multi-centre randomized controlled trial. Acupunct Med. 2023 Apr;41(2):86-95. doi: 10.1177/09645284221086289. Epub 2022 Jun 7. PMID 35673804